CLINICAL TRIAL: NCT00986492
Title: Influence de la Privation Aigue de Sommeil Sur la Prise Alimentaire et l'activité Physique Chez l'Homme
Brief Title: Effects of Sleep Deprivation on Food Intake and Motor Activity in Man
Status: Completed | Type: Observational
Sponsor: University Hospital, Caen (Other)
Collaborators: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Pr Pierre Denise, University Hospital, Caen
Other Study IDs: 2009-A00297-50
Record Dates: First submitted 2009-09-24; First posted 2009-09-30 (Estimated); Last update posted 2009-09-30 (Estimated); Status verified 2009-09

CONDITIONS: Healthy
Keywords: Sleep deprivation; Food intake; Motor activity; Normal, healthy subjects
MeSH Terms: conditions — Sleep Deprivation; Motor Activity

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Evidence that shortened period of sleep could be a risk factor for weight gain and obesity has grown over the past decade. Concurrent with the obesity epidemic, numerous studies have reported a parallel epidemic of chronic sleep deprivation. Sleep is important in maintaining energy balance (i.e. acute sleep deprivation impact the normal secretion of ghrelin and decreases leptin plasma levels). Surprisingly, in humans, there is no direct evidence that a shortened night has direct effect on energy metabolism during the following day.

This study is set up to determine whether a partial sleep deprivation night has an impact on appetite and food energy intake and, concomitantly, on physical activity, during the following day.

ELIGIBILITY:
Inclusion Criteria:

* male
* age between 18 and 30
* healthy
* non smoker
* less than 5 hour of sport per week
* BMI between 20 and 25 kg/m/m

Exclusion Criteria:

* eating disorders,
* dieting or fasting
* restrained (score >9), disinhibited (score >11) or hungry subjects (score >9), according to the Three-Factor Eating Questionnaire general healthiness,
* food-snacking (more than twice a day),

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy normal subjects
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2009-04; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Daily food intake | 24h

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Denise, MD, PhD, Principal Investigator — University Hospital, Caen

REFERENCES:
- [Derived] Brondel L, Romer MA, Nougues PM, Touyarou P, Davenne D. Acute partial sleep deprivation increases food intake in healthy men. Am J Clin Nutr. 2010 Jun;91(6):1550-9. doi: 10.3945/ajcn.2009.28523. Epub 2010 Mar 31. PMID 20357041